CLINICAL TRIAL: NCT03768960
Title: A Prospective, Single-Arm, Multicenter, Pragmatic Phase-IV Trial Investigating Safety and Effectiveness of DARZALEX (Daratumumab) In Indian Subjects With Relapsed and Refractory Multiple Myeloma, Whose Prior Therapy Included a Proteasome Inhibitor and an Immunomodulatory Agent
Brief Title: A Study of DARZALEX (Daratumumab) In Indian Participants With Relapsed and Refractory Multiple Myeloma, Whose Prior Therapy Included a Proteasome Inhibitor and an Immunomodulatory Agent
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Johnson & Johnson Private Limited (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CR108556; 54767414MMY4008 (Other: Johnson & Johnson Private Limited)
Record Dates: First submitted 2018-11-29; First posted 2018-12-07 (Actual); Last update posted 2025-02-03 (Actual); Status verified 2025-01

CONDITIONS: Multiple Myeloma
MeSH Terms: conditions — Multiple Myeloma | interventions — daratumumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Daratumumab (Experimental): Participants will receive 16 milligram per kilogram (mg/kg) of daratumumab as intravenous (IV) infusion every week (QW) in Cycles 1 and 2 (Days 1, 8, 15 and 22) and every 2 weeks (Q2W) in Cycle 3 to 6 (Days 1 and 15) each cycle is of 28 days.
  Interventions: Drug: Daratumumab

INTERVENTIONS:
Drug: Daratumumab — Participants will receive 16 mg/kg of daratumumab as IV infusion QW in Cycles 1 and 2 (Days 1, 8, 15 and 22) and Q2W in Cycle 3 to 6 (Days 1 and 15).
  Other Names: DARZALEX

SUMMARY:
The purpose of this study is to demonstrate the safety profile of daratumumab in routine clinical practice when given as monotherapy in Indian participants with relapsed and refractory multiple myeloma, whose prior therapy included a proteasome inhibitor and an immunomodulatory agent.

ELIGIBILITY:
Inclusion Criteria:

* Participants with relapsed and refractory multiple myeloma (as per International Myeloma Working Group [IMWG] definitions) whose prior therapy included a proteasome inhibitor and an immunomodulatory agent, being newly initiated on DARZALEX (daratumumab) monotherapy based on independent clinical judgment of treating physicians as per locally approved prescribing information
* Each participant (or their legally acceptable representative) must sign an informed consent form (ICF) indicating that he or she understands the purpose of and procedures required for the study and are willing to participate in the study. Participants must be willing and able to adhere to the prohibitions and restrictions specified in this protocol, as referenced in the informed consent form (ICF)

Exclusion Criteria:

* Participants who are not eligible to receive DARZALEX as per the locally approved prescribing information
* Participant participating or planning to participate in any interventional drug trial during the course of this study
* Known seropositive for human immunodeficiency virus (HIV)
* Seropositive for hepatitis B (defined by a positive test for hepatitis B surface antigen [HBsAg]). Participants with resolved infection (that is, participants who are HBsAg negative but positive for antibodies to hepatitis B core antigen [anti-HBc] and/or antibodies to hepatitis B surface antigen [anti-HBs]) must be screened using real-time polymerase chain reaction (PCR) measurement of hepatitis B virus (HBV) deoxyribonucleic acid (DNA) levels. Those who are PCR positive will be excluded. exception: Participants with serologic findings suggestive of HBV vaccination (anti-HBs positivity as the only serologic marker) and a known history of prior HBV vaccination, do not need to be tested for HBV DNA by PCR
* Known seropositive for hepatitis C (except in the setting of a sustained virologic response [SVR], defined as aviremia at least 12 weeks after completion of antiviral therapy)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Actual)
Dates: Start 2019-06-10 (Actual); Primary Completion 2022-07-16 (Actual); Study Completion 2022-07-16 (Actual)

PRIMARY OUTCOMES:
Incidence of Treatment Emergent Adverse Events (TEAE) | Approximately up to 29 weeks
  An adverse event (AE) is any untoward medical occurrence attributed to study drug in a participant who received study drug.

SECONDARY OUTCOMES:
Overall Response Rate (ORR) | Approximately up to 24 weeks
  ORR- % of participants who achieve partial response (PR) or better per IMWG criteria during study treatment. PR: >=50% reduction of serum M-protein, >=90% reduction in 24 hour urinary M-protein or to<200mg/24hour; if serum and urine M-protein are not measurable, >=50% decrease in difference between involved and uninvolved free light chain (FLC) level; if serum and urine M-protein and serum free light assay is not measurable, >=50% reduction in bone marrow plasma cell (PC), with baseline bone marrow PC% >=30%; if present at baseline, >=50% reduction in size of soft tissue plasmacytomas; VGPR: serum and urine M-component detectable by immunofixation or >=90% reduction in serum M-protein and urine M-protein <100mg/24hour; Complete response(CR):negative immunofixation on serum and urine, disappearance of soft tissue plasmacytomas and <5% PCs in bone marrow; sCR: CR and normal FLC ratio, absence of clonal PCs by immunohistochemistry, immunofluorescence or 2 to 4 color flow cytometry.
Percentage of Participants with Very Good Partial Response (VGPR) or better | Approximately up to 24 weeks
  VGPR or better is defined as percentage (%) of participants with a response of very good partial response (VGPR) or better according to the International Myeloma Working Group (IMWG) criteria, during the study treatment. IMWG criteria for VGPR: serum and urine M-component detectable by immunofixation or greater than or equal to (>=)90% reduction in serum M-protein and urine M-protein less than (<)100 milligram(mg)/24hour; CR: Negative immunofixation on the serum and urine, disappearance of any soft tissue plasmacytomas, and <5% PCs in bone marrow; Stringent CR (sCR): CR and normal FLC ratio, absence of clonal PCs by immunohistochemistry, immunofluorescence or 2 to 4 color flow cytometry.
Percentage of Participants with Progression Free Survival (PFS) | Approximately up to 24 weeks
  PFS is defined as % of participants with PFS from date of randomization to either PD, according to the IMWG criteria or death, whichever occurs first. PD: Increase of >=25% in level of serum M-protein from lowest response value and absolute increase must be >=0.5 gram per deciliter (g/dL); Increase of >=25% in 24 hours urinary light chain excretion (urine M-protein) from lowest response value and absolute increase must be >=200 mg/24 hour; Only in participants without measurable serum and urine M-protein levels: increase of >=25% in difference between involved and uninvolved FLC levels from lowest response value and absolute increase must be greater than (>)10 milligram per deciliter (mg/dL); Definite increase in size of existing bone lesions or soft tissue plasmacytomas; Definite development of new bone lesions or soft tissue plasmacytomas; Development of hypercalcemia (corrected serum calcium >11.5 mg/dL) that can be attributed solely to PC proliferative disorder.
Time to Response | Approximately up to 24 weeks
  Time to Response: time between the date of randomization and the first effectiveness evaluation that the participant has met all criteria for CR or PR. CR: negative immunofixation on serum and urine, disappearance of soft tissue plasmacytomas and <5% PCs in bone marrow; PR: greater than or equal to (>=) 50% reduction of serum M-protein, >=90% reduction in 24 hour urinary M-protein or to less than (<) 200 mg/24 hours; if serum and urine M-protein are not measurable, >=50% decrease in difference between involved and uninvolved free light chains (FLC) levels; if serum and urine M-protein and serum free light assay is not measurable, >=50% reduction in bone marrow plasma cell (PC), with baseline bone marrow PC percentage >=30%; if present at baseline, >=50% reduction in size of soft tissue plasmacytomas.
Change from Baseline in European Organization for Research and Treatment of Cancer Quality of Life Questionnaire (EORTC QLQ-C30) Score | Baseline, Day 1 (Cycle 1 to 5); Days 1 and 28 (Cycle 6) (each cycle of 28 days)
  The EORTC QLQ-C30 is a 30-item questionnaire containing both single and multi-item measures. These include five functional scales (Physical, Role, Cognitive, Emotional, and Social Functioning), three symptom scales (Fatigue, Pain, and Nausea/Vomiting), a Global Health Status/ Quality-of-Life (QoL) scale, and six single items (Constipation, Diarrhea, Insomnia, Dyspnea, Appetite Loss, and Financial Difficulties). The scores ranges from 0-100, a high score for functional scales and for Global Health Status/QoL represent better functioning ability or Health-Related Quality-of-Life (HRQoL), whereas a high score for symptom scales and single items represents significant symptomatology.
Change from Baseline in EuroQol-5 Dimensions (EQ-5D-5L) Score | Baseline, Day 1 (Cycle 1 to 5); Days 1 and 28 (Cycle 6) (each cycle of 28 days)
  EQ-5D-5L is a 5-item questionnaire that assesses 5 domains including mobility, self-care, usual activities, pain/discomfort and anxiety/depression plus a visual analog scale rating "health today" with ranges from 0 (worst imaginable health state) to 100 (best imaginable health state). Each dimension has 5 response options (no problems, slight problems, moderate problems, severe problems and extreme problems) that reflect increasing levels of difficulty. The responses to the 5 dimensions are used to compute a single utility score ranging from zero (0.0- worst health state) to 1 (1.0- better health state) representing the general health status of the individual.

CONTACTS AND LOCATIONS:
Overall Officials: Johnson & Johnson Private Limited Clinical Trial, Study Director — Johnson & Johnson Private Limited
Locations (16):
- India (16):
  - Avron Hospitals Pvt. Ltd, Ahmedabad
  - M S Ramaiah Medical College and Hospital, Bengaluru
  - Sparsh Hospitals & Critical Care (Pvt) Ltd, Bhubaneshwar
  - Apollo Hospitals, Bhubaneswar
  - Post Graduate Institute of Medical Education And Research PGIMER, Chandigarh
  - Apollo Hospitals, Hyderabad
  - Basavatarakam Indo-American Hospital, Hyderabad
  - Cytecare Hospitals Pvt. Ltd, Karnataka
  - Tata Medical Center, Kolkata
  - Shatabdi Super Speciality Hospital, Mumbai Naka
  - Kingsway Hospital, Nagpur
  - Apex Wellness Hospital, Nashik
  - All India Institute of Medical Sciences, New Delhi
  - Jawaharlal Institute of Postgraduate Medical Education and Research, Puducherry
  - Deenanath Mangeshkar Hospital and Research Centre, Pune
  - Noble Hospital Pvt Ltd, Pune

REFERENCES:
- [Derived] Kumar L, Melinkeri S, Ganesan P, Kumar J, Biswas G, Kilara N, Pathalingappa H, Prasad S, Jain M, Mishra SK, Prasad S, Boyella PK, Sahoo RK, Bondarde S, Shah S, Rege M, Deb U, Korde T, Dixit J. Daratumumab in Indian patients with relapsed and refractory multiple myeloma: a prospective, multicenter, phase IV study. Future Oncol. 2024 Feb;20(4):191-205. doi: 10.2217/fon-2023-0842. Epub 2023 Dec 20. PMID 38116642